CLINICAL TRIAL: NCT03612518
Title: An mHealth, Multi-Centre Randomized Controlled Trial to Promote Use of Postpartum Contraception Amongst Rural Women in Punjab, Pakistan
Brief Title: An mHealth Trial to Promote the Use of Postpartum Contraception
Acronym: PPFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Junaid-ur-Rehman Siddiqui (Other)
Responsible Party: Sponsor-Investigator, Junaid-ur-Rehman Siddiqui, Principal Investigator, Marie Stopes Society
Organization: Marie Stopes Society (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 009-17
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Contraception Behavior
Keywords: postpartum family planning; RCT; mhealth
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text and Voice Messages (Experimental): Participants will receive text messages and voice messages
  Interventions: Behavioral: Text and Voice Messages
- Interactive Phone Call (Experimental): Participants will receive interactive phone calls
  Interventions: Behavioral: Interactive Phone Call
- Control (No Intervention): Participants in this arm will not be exposed to any intervention.

INTERVENTIONS:
Behavioral: Text and Voice Messages — Participants in this study arm will periodically receive information regarding antenatal- and postnatal care and family planning services through text and voice messages from the fifth gestational month until the post-partum period of 42 days.
  Arms: Text and Voice Messages
Behavioral: Interactive Phone Call — Participants in this study arm will receive information regarding antenatal- and postnatal care and family planning services through periodic interactive phone calls from the fifth gestational month until the post-partum period.
  Arms: Interactive Phone Call

SUMMARY:
Multiple encounters of pregnant women with the health care system during the late antenatal and immediate postpartum period provide a gateway for postpartum family planning counselling. Counselling on family planning services during this time is considered effective and cost-efficient for promoting healthy timing and spacing of pregnancies. This research aims to test the effectiveness of mobile phone-based interventions in promoting use of postpartum contraception.

DETAILED DESCRIPTION:
The study will be a three-arm, 10-month, multicentre, parallel-group, randomized controlled trial which will be conducted at 15 Suraj social franchise(SF) health facilities in Punjab province of Pakistan. Pregnant women aged 15-44 years who are in their first or second trimester and have a mobile phone for their own use will be eligible to participate in this study. The participants will be randomly allocated to one of three study arms: a) voice and text messages; b) interactive telephone-based counselling; or c) control arm (no additional phone-based support). The intervention counselling module will be developed based on the Integrated Behaviour Model which was recently adapted, and tested for the family planning context in Pakistan. It will broadly cover birth-preparedness, birth spacing and contraception, and postnatal care. The phone-based intervention aims to improve women's ability to use contraception by providing them with information about a range of methods, access to family planning methods through outlets such as Suraj SF providers, connecting them with MSS field health educators to help them reach the centres, motivation by re-enforcing the benefits of contraceptive use on women's quality of life, and dispelling myths and misconceptions about modern contraceptive methods. Risk differences will be used as the measure of effect of the intervention on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Married
* Pregnant women with gestational age up to 20 weeks
* 15-44 years old throughout duration of study
* Literate
* Access to a cellphone
* Living in the study's catchment area

Exclusion Criteria:

* Not up to 20 weeks pregnant
* Not between 15-44 years old for the study duration
* Illiterate
* Does not have regular access to a cellphone
* Not residing within the catchment area
* Does not provide consent to participate

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 970 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Contraceptive Uptake | Through study completion, an average of six months
  Proportion of subjects enrolled in each of the three groups who adopt any modern family planning method to delay next pregnancy
Skilled Birth | Through study completion, an average of six months
  Proportion of women who gave birth in a health facility or through a skilled birth professional
Immunisation | Through study completion, an average of six months
  Proportion of women reported to immunise the newborn at birth

SECONDARY OUTCOMES:
Intention to Adopt Modern Contraception | Through study completion, an average of six months
  The proportion of subjects enrolled in the program who state that they intend to adopt any modern family planning method to delay their next birth by 24 months (by type contraceptive method and time within 42 days of postpartum period)

CONTACTS AND LOCATIONS:
Overall Officials: Xaher Gul, DrPH(c), Principal Investigator — Marie Stopes Society; Waqas Hameed, MSc, Principal Investigator — Marie Stopes Society; Junaid-ur-Rehman Siddiqui, BBA, Principal Investigator — Marie Stopes Society; Sharmeen Hussain, MPH, Principal Investigator — Marie Stopes Society; Ishaque Sheikh, MSc, Principal Investigator — Marie Stopes Society
Locations (4):
- Pakistan (4):
  - Suraj Social Franchise, Hafizabad, Punjab Province
  - Suraj Social Franchise, Jhang, Punjab Province
  - Suraj Social Franchise, Kasur, Punjab Province
  - Suraj Social Franchise, Toba Tek Singh, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
IPD will only be shared for underlying results in a publication. Furthermore, de-identified participant data pertinent only to the research paper will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Publication
Access Criteria: At the time of publication, data will be submitted to a data repository and the URL will be shared with the journal, and the journal will make the information public. Requests to access data will be individually reviewed by the research team.

REFERENCES:
- [Background] Smith C, Gold J, Ngo TD, Sumpter C, Free C. Mobile phone-based interventions for improving contraception use. Cochrane Database Syst Rev. 2015 Jun 26;2015(6):CD011159. doi: 10.1002/14651858.CD011159.pub2. PMID 26115146
- [Background] Cleland J, Shah IH, Daniele M. Interventions to Improve Postpartum Family Planning in Low- and Middle-Income Countries: Program Implications and Research Priorities. Stud Fam Plann. 2015 Dec;46(4):423-41. doi: 10.1111/j.1728-4465.2015.00041.x. PMID 26643491
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Gul X, Hameed W, Hussain S, Sheikh I, Siddiqui JU. A study protocol for an mHealth, multi-centre randomized control trial to promote use of postpartum contraception amongst rural women in Punjab, Pakistan. BMC Pregnancy Childbirth. 2019 Aug 8;19(1):283. doi: 10.1186/s12884-019-2427-z. PMID 31395034